CLINICAL TRIAL: NCT06802146
Title: A Multi-Site Break Through Cancer Pilot Study Testing the Feasibility and Safety of Therapeutic Intervention for Patients With High-risk Clonal Cytopenia of Undetermined Significance (CCUS)
Brief Title: Early Intervention in High Risk CCUS
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Lachelle D. Weeks, MD, PhD (Other)
Collaborators: Astex Pharmaceuticals, Inc. (Industry); Break Through Cancer (Unknown)
Responsible Party: Sponsor-Investigator, Lachelle D. Weeks, MD, PhD, Sponsor-Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-658
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Clonal Cytopenia of Undetermined Significance; Cytopenia
Keywords: Clonal Cytopenia of Undetermined Significance; CCUS; Cytopenia
MeSH Terms: conditions — Cytopenia | interventions — decitabine and cedazuridine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inqovi Cohort (Experimental): Participants will be enrolled and will complete:
  * Baseline visit.
  * In-clinic visits with assessments: Cycle 1 days 8, 15, and 22.
  * In-clinic visits with assessments and bone marrow biopsies: Cycles 2 - 12 Day 1.
  * Cycle 1 - 12:
    • Days 1 - 5 of 28 day cycle: Predetermined dose of Inqovi 1x daily.
  * End of Treatment visit, Cycle 13 Day 1, with assessments and bone marrow biopsy.
  * Follow up in-clinic visits with assessments: Cycle 19 Day 21, Cycle 25 Day 1, Cycle 31 Day 1, and Cycle 36 Day 28. Bone marrow biopsy at Cycle 25 Day 1.
  * End of Study visit, Cycle 36 Day 28, with assessments and bone marrow biopsy.
  Interventions: Drug: Inqovi
- Observational Cohort (No Intervention): Participants will complete:
  * Baseline visit.
  * In-clinic visits with assessments: Cycle 7 Day 1, Cycle 13 Day, Cycle 19 Day, Cycle 25 Day 1, and Cycle 31 Day 1.
  * Bone marrow biopsies every 12 months at Cycle 13 Day 1 and Cycle 25 Day.
  * End of study visit, Cycle 36 Day 28, with assessments and bone marrow biopsy.

INTERVENTIONS:
Drug: Inqovi — Combination of a nucleoside metabolic inhibitor and cytidine deaminase inhibitor, 10mg DEC / 100mg CED tablet, taken orally per protocol.
  Other Names: Decitabine and Cedazuridine; ASTX727
  Arms: Inqovi Cohort

SUMMARY:
This research is being done to find out more about the potential risks and benefits of early treatment in participants with high risk Clonal Cytopenia of Unknown Significance (CCUS). This study will give eligible CCUS participants the option of either being observed or taking an oral drug as treatment.

The names of the study drug involved in this study is:

-Decitabine/cedazuridine (DEC/CED) (a nucleoside metabolic inhibitor and cytidine deaminase inhibitor).

DETAILED DESCRIPTION:
This is an open-label, multicenter pilot study testing the feasibility and safety of early pharmacologic intervention, decitabine/cedazuridine, in participants with higher-risk clonal cytopenia of unknown significance (CCUS).

The U.S. Food and Drug Administration (FDA) has not approved DEC/CED for CCUS but it has been approved for other uses.

The research study procedures include screening for eligibility, in-clinic treatment visits, electrocardiograms, echocardiograms, bone marrow biopsies, and blood tests.

Participants who choose to enroll in the intervention cohort will receive the oral drug for 1 year and will continue in a post-treatment observation period for 2 years after treatment. Participants in both groups will each participate in the study for 3 years total.

It is expected that the study will continue to enroll up to 108 participants in total or until there are 30 participants enrolled in the early intervention cohort, whichever occurs first.

Astex Oncology is funding this research study by providing the drug Decitabine/cedazuridine.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Unexplained cytopenia(s) for at least 4 months (at least two separate labs within 4 months including at time of screening must meet this criteria). Cytopenia(s) defined as the presence of ≥ 1 of the following:

  * Hemoglobin (Hgb) <12 g/dL for women and <13g/dL for men
  * Absolute neutrophil count (ANC) < 1.8 × 109/L*
  * Platelet count (Plt) <150 × 109/L *Patients known to have a Duffy-null genotype must have anemia (Hgb < 12g/dL for women, Hgb <13g/dL for men) and/or thrombocytopenia (Plt < 150 × 109/L) to be eligible for this study.

    * 1 pathogenic variant detected in any myeloid driver gene with a VAF of at least 0.02 (2%) identified by local next generation sequencing (NGS) of peripheral blood or bone marrow sample within 3 months from screening bone marrow biopsy.
* Participants must have a high risk score per the Clonal Hematopoiesis Risk Calculator (CHRS). See APPENDIX C for calculation.
* Screening bone marrow biopsy must not be diagnostic of any overt hematologic malignancy by morphologic assessment and must be consistent with a diagnosis of clonal cytopenia of unknown significance (CCUS) as determined by multi-institutional hematopathology review.
* ECOG performance status 0-2 (see Appendix A).
* Participants must meet the following organ function as defined below:

  * Serum aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤3x upper limit of normal (ULN).
  * Serum total bilirubin <1.5x ULN. Higher levels are acceptable if these can be attributed to ineffective erythropoiesis or Gilbert's syndrome. In these cases, approval from the study Sponsor-Investigator is required.
  * Creatinine clearance greater than 40 mL/min based on the Cockcroft-Gault glomerular filtration rate estimation.
* Ability to understand and the willingness to sign a written informed consent document.
* For participants of the early pharmacologic intervention cohort: women of childbearing potential must use highly effective contraception during treatment for at least 6 months after the last dose and males with female partners of reproductive potential should use effective contraception during treatment and for 3 months after the last dose.

Exclusion Criteria:

* Concurrent primary malignancy requiring active cytotoxic chemotherapy and/or ionizing radiation therapy.
* Known inherited bone marrow failure disorder and/or germline predisposition to hematologic malignancy.
* Receipt of anti-cancer therapy including any cytotoxic chemotherapy, ionizing radiation therapy, immunomodulatory agents such as lenalidomide, and targeted anti-cancer therapies including PARP inhibitors within the last 6 months. Patients with complete surgical resection of a tumor are not excluded from this study.
* Anti-cancer therapy, including any cytotoxic chemotherapy, ionizing radiation therapy, immunomodulatory agents such as lenalidomide and targeted agents such as PARP inhibitors, planned in the next 6 months. Patients on hormonal adjuvant therapy for nonmetastatic breast and prostate cancer or other minimally-myelosuppressive maintenance therapies for non-metastatic cancer may be eligible at the discretion of the study PI.
* Diagnosis of MDS, MPN, CMML, AML or any other hematolymphoid malignancy in the patient's lifetime. This includes individuals with MDS-defining chromosomal abnormalities identified via conventional karyotype or FISH.
* Presence of a concurrent hematologic malignancy precursor state, such as smoldering multiple myeloma (SMM), and smoldering Waldenstrom's macroglobulinemia.
* Presence of an early-stage hematologic precursor state-such as monoclonal gammopathy of undetermined significance (MGUS) and monoclonal B cell lymphocytosis (MBL).
* Active uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment).
* Recent (within 3 months) vaccination with any live attenuated vaccine or vaccination with live attenuated vaccine planned during the next 15 months. *Live attenuated vaccines include measles, mumps, rubella (MMR combined vaccine), rotavirus, smallpox, chickenpox, and yellow fever.
* Laboratory evidence indicative of clinically significant red cell hemolysis.
* Hypersplenism and/or evidence of portal hypertension on physical exam or imaging.
* Pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility Failure Rate (FFR) | Treatment duration up to 12 cycles (28 days per cycle).
  FFR is defined by the proportion of eligible subjects with higher risk CCUS who enter the study and opt to participate in the early intervention as opposed to observation only cohort.

SECONDARY OUTCOMES:
Grade 3-5 Treatment-related Toxicity Rate | AE evaluated on treatment at day 1, 8, 15, 22 on cycle 1, then day 1 on cycle 2-12, and EOT. Median treatment duration for this study cohort was 6 months (range T1- T2).
  All grade 3-5 adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv5 that are not resolved in accordance with treatment guidelines were counted. Rate is the percentage of treated participants experiencing at least one of these adverse events as defined during the time of observation.
Treatment Tolerability Rate (TTR) | Treatment up to 12 cycles, (28 days per cycle).
  TTR will be measured by the percentage of participants in the early intervention treatment arm that complete ≥3 cycles of oral DEC/CED.
Hematologic Response Rate (HRR) | Response collected every 3 months on treatment. Treatment duration up to 12 cycles, (28 days per cycle).
  HRR defined as proportion of participants achieved hematologic response by 2018 World Health Organization (WHO) International Working Group (IWG) MDS response criteria.
Median Overt Myeloid Neoplasia (MN)-Free Survival | Disease evaluated every 3 months on treatment, then every 12 months off treatment, up to 2 years for interventional cohort, up to 3 years for observation cohort.
  MN-free survival based on the Kaplan-Meier method is defined as the duration of time from study entry to overt myeloid neoplasia diagnosed per the 5th edition of the WHO Classification of Haematolymphoid Tumors.
Somatic Driver Mutation Variant Allele Frequencies (VAFs) Reduction Rate | Clinical next generation sequencing (NGS) is collected every 3 month on treatment, for up to 12 cycles, (28 days per cycle).
  Changes in variant allele fraction (VAF) will be assessed as a biomarker for clone size. A clinically significant VAF reduction will be defined as a persistent (evident on 2 sequential measurements 3 or more months apart) VAF reduction of the pathogenic mutation in question of ≥10%, or for initial VAFs <10%, if the mutation becomes undetectable. Rate defines as proportion of participants achieved the VAFs reduction.
Changes in Serum Inflammatory Markers | High sensitivity CRP will be measured at screening, every 6 months, and at end of study/disease progression, up to 3 years.
  Serum Inflammatory Markers measured using established method. Change will be defined as percentage increase/decrease from baseline measurement at screening.
Change in Score of the Adult Comorbidity Evaluation 27 (ACE-27) | Survey is evaluated at screening, every 6 months, and at end of study/disease progression, up to 3 years.
  Adult Comorbidity Evaluation-27 identify the important medical comorbidities and grade severity using the index. Overall Comorbidity Score is defined according to the highest ranked single ailment, except in the case where two or more Grade 2 ailments occur in different organ systems. In this situation, the overall comorbidity score should be designated Grade 3. Overall score range from 0-None to 3-Serve, and noted 9-Unknown.
Change in Score of the 36-item Short Form Survey (SF-36) | Survey is evaluated at screening, every 6 months, and at end of study/disease progression, up to 3 years.
  The Short Form (SF)-36 is a 36-item participant-reported questionnaire that covers eight health domains. Scores for each domain range from 0 to 100%. To score the SF-36, scales are standardized with a scoring algorithm or by SF-36 scoring software to obtain a score ranging from 0 to 100. Higher scores indicate better health status, and a mean score of 50 has been articulated as a normative value for all scales.

CONTACTS AND LOCATIONS:
Overall Officials: Lachelle Weeks, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu